CLINICAL TRIAL: NCT05341544
Title: Non-invasive Vagal Stimulation for Frequent Premature Ventricular Complexes (NoVa-PVC)
Brief Title: Non-invasive Vagal Stimulation for Frequent Premature Ventricular Complexes
Acronym: (NoVa-PVC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Stavros E Mountantonakis, Director, Cardiac Electrophysiology, Lenox Hill Hospital, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-0076
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Premature Ventricular Contraction
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to either LLTS first and then sham-stimulation, or sham-stimulation first and then LLTS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Patients will receive 1 hour of active low level tragus stimulation daily for 10 days.
  Interventions: Device: Parasym device
- Sham (Sham Comparator): Patients will receive 1 hour of sham low level tragus stimulation daily for 10 days.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Parasym device — The study will utilize the Parasym device (Parasym Health, London, United Kingdom) paired with compatible electrodes to administer the transcutaneous LLTS.
  Arms: Active
Device: Sham device — Sham device
  Arms: Sham

SUMMARY:
A prospective sham-controlled randomized clinical trial to assess the effect of low-level tragus stimulation (LLTS) in patients with frequent premature ventricular complexes (PVCs)

DETAILED DESCRIPTION:
This is a two-center, prospective, cross-over, sham-controlled, double-blinded, randomized clinical trial. All the patients will receive a cardiac event monitor at baseline for 28 days, the patient will switch the ePatch after 14 days . Patients will be allocated to either LLTS first and then sham-stimulation, or sham-stimulation first and then LLTS. Each treatment period (sham-stimulation and LLTS) will last 10 days. The Parasym device will be used, and the patients will receive LLTS or sham-stimulation for 1 hour daily. The wash-out period between the two treatments will last 8 days. Patients will be continually monitored via event monitor for 28 days in duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old) but < 80 years of age
* Symptomatic PVCs or asymptomatic PVCs with a burden > 5%
* Intolerant to or unwilling to take beta blockers and nondihydropyridine calcium channel blockers or beta blockers and nondihydropyridine calcium channel blockers have proved ineffective

Exclusion Criteria:

* Ischemic cardiomyopathy with LVEF < 40%
* Severe heart failure (New York Heart Association Class III, or IV) or valve disease
* Sustained ventricular tachycardia
* Structural heart disease or myocardial scar
* Pregnancy or nursing
* Patients with known thyroid issues, on renal dialysis.
* Patients with prolonged first-degree block, high degree AV block (2nd or 3rd degree), bivascular block and documented sick sinus syndrome
* Hypotension due to autonomic dysfunction
* Patients with cardiac implantable electronic device (ICD or PPM) , hearing aid implants or any implanted metallic or electronic device
* Patients who have had prior cervical vagotomy
* Patients with skin on the tragus that is broken or cracked
* Patients with a history of baseline cardiac disease or atherosclerotic cardiovascular disease, including congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction (within 5 years) and patients diagnosed with narrowing of the arteries (carotid atherosclerosis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
PVC Burden | 28 days
  Daily PVC Count by event monitor

SECONDARY OUTCOMES:
Quality of life survey | 28 days
  SF 36 QOL Score
Heart Rate Variability | 28 days
  Daily HRV
PVC Morphology | 28 days
  Fluctuation in PVC Morphology by event monitor

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwell Health, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zafeiropoulos S, Coleman K, Kogan J, Varrias D, Leavitt J, Bekiaridou A, Zanos T, Zanos S, Stavrakis S, Mountantonakis S. Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Premature Ventricular Contractions: A Crossover, Randomized Clinical Trial (NoVa-PVC). JACC Clin Electrophysiol. 2025 Aug;11(8):1699-1707. doi: 10.1016/j.jacep.2025.04.011. Epub 2025 Apr 24. PMID 40392172